CLINICAL TRIAL: NCT04010136
Title: Identification of Elderly Patients in Need of Palliative Care by Family Physicians - the Role of Palliative Care Training and the Use of a Standardized Tool (GerPal_ID). A Two-phase Protocol: Randomized Trial and Prevalence Study
Brief Title: Identification of Elderly Patients in Need of Palliative Care by Family Physicians
Acronym: GerPal-ID
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We were not able to recruit participants to enrol the study. As it was not able, the investigation team decided not to proced.
Sponsor: University of Beira Interior (Other)
Responsible Party: Principal Investigator, Carlos Seiça Cardoso, Principal Investigator, University of Beira Interior
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CE-UBI-Pj-2019-023:ID1244
Record Dates: First submitted 2019-06-14; First posted 2019-07-08 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Palliative Care; Primary Health Care; Geriatrics
Keywords: Palliative care; Primary health care; Palliative care training; Prevalence; Geriatrics

STUDY DESIGN:
Intervention Model Description: The GPs (fellows and specialists) from Center Healthcare Administrative Region will be invited to take part in this trial. The invitations will be conducted with the help of the Center Healthcare Administrative Region and by spreading the invitation in some general practice professionals' mailing lists and online platforms.
  First, GPs will be contacted and those who accept to participate will be randomized into one of the four-harm study groups - 1. Control Group, 2. Identification tool group, 3. Standard PC training, 4 - Clinical cases based PC training.
  The accuracy on the identification before and after intervention will be compared within each group and between the four groups using a clinical record based identification tool (CCB-PCId).
  A PC expert panel will build a tool, clinical record based, to evaluate the accuracy of palliative care needs identification.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): GPs (fellows and specialists) from Center Healthcare Administrative Region that will be given no intervention
- Identification tool group (Experimental): GPs (fellows and specialists) from Center Healthcare Administrative Region that will receive access to the Identification tool Supportive and Palliative Care Indicators Tool (SPICT-PT) with a brief training on how to use it.
  Interventions: Other: Palliative care training
- Standard Palliative Care Training (Experimental): GPs (fellows and specialists) from Center Healthcare Administrative Region that will receive palliative care training according to the Center Healthcare Administrative Region standard model of training.
  Interventions: Other: Palliative care training
- Clinical cases based Palliative Care Training (Experimental): GPs (fellows and specialists) from Center Healthcare Administrative Region that will receive palliative care training using a clinical cases based model.
  Interventions: Other: Palliative care training

INTERVENTIONS:
Other: Palliative care training — Intervention will consist on providing different types of palliative care training to identify the most accurate on improving GPs' identification of palliative care patients skills
  Arms: Clinical cases based Palliative Care Training; Identification tool group; Standard Palliative Care Training

SUMMARY:
In the last decades, the number of people living with chronic diseases had increased, mainly due to the aging of the population. Such chronic, progressive, life threatening and burdening diseases, play an important role in this new era of palliative care.

Despite the growing scientific and social interest in palliative care, there is still a delay in the identification of patients with palliative care needs. This leads to a late integration in a palliative care network and consequent deprivation of the major advantages of an early and progressive integration.

The aim of this study is to evaluate the role of palliative care training and the use of a structured tool, in the identification of the elderly population in need of palliative care by family physicians. And also to conduct a prevalence study to further the knowledge about how many elder people in primary care have the need of a palliative care approach.

DETAILED DESCRIPTION:
The study consists of two phases:

1. Randomized trial with General Practitioners (GP) to determine the role of two different training programs and a structured tool in the identification of geriatric patients with palliative care needs.
2. Cross-sectional, analytical study of the prevalence and patterns of geriatric patients with Palliative Care (PC) needs, managed in primary care in Portugal's Center Healthcare Administrative Region.

ELIGIBILITY:
Inclusion Criteria:

* GPs (fellows and specialists) from Center Healthcare Administrative Region

Exclusion Criteria:

* Previous palliative care training.
* Refuse to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-12-29 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
GPs' rate of identification of patients with palliative care needs | 2 weeks
  Each GP will have to identify, before each intervention, from a set of fictitious clinical cases constructed for this purpose, which patients need palliative care. After each intervention, they will re-evaluate the same clinical cases and will be asked to identify again which patients need palliative care.
  Each intervention will be measured according to the identification accuracy.
Prevalence geriatric patients with palliative care needs | 6 months
  Number (% of patients) of geriatric patients, managed in primary care in Center Healthcare Administrative Region, with palliative care needs.
Sociodemographic characteristics of geriatric patients with palliative care needs | 6 months
  Age (in years), sex (male or female), marital status (single, married, divorced, widow, marriage) and job of geriatric patients, managed in primary care in Center Healthcare Administrative Region, with palliative care needs.
Clinical characteristics of geriatric patients with palliative care need | 6 months
  Main diseases, main symptoms, number of contacts with GP/year of geriatric patients, managed in primary care in Center Healthcare Administrative Region, with palliative care needs.
Complexity of geriatric patients with palliative care need | 6 months
  Complexity of of geriatric patients, managed in primary care in Center Healthcare Administrative Region, with palliative care needs, evaluated using ICD-Pal tool

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Seiça Cardoso, MD, Principal Investigator — Faculty of Health Science - University of Beira Interior
Locations (1):
- Center Healthcare Administrative Region, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Yes
The study will be conducted in accordance with the principles expressed in the Declaration of Helsinki. It has full approval from the Ethics Committee of the Faculty of Health Sciences, University of Beira Interior. Study results will be published in peer-reviewed journals and presented at national and international conferences.
Supporting Information: Study Protocol, CSR
Time Frame: Between June 2019 and October 2020
Access Criteria: A descriptive analysis will be performed to all study variables, namely the number of valid observations, mean, standard deviation, median and range for quantitative variables and absolute and relative frequencies for qualitative variables whenever it will be considered adequate.
  According to previous reports , patients with palliative care needs will be defined as ≥2 positive general indicators or ≥1 positive disease-specific indicators in the SPICT.
  Comparisons between two or more independent groups of quantitative variables will be performed using Pearson's Chi2 test or Fisher's exact test, analysis of variance (ANOVA) or non-parametric Kruskal-Wallis test. All tests will be two-sided using a significance level of 0.05. Statistical analysis will be conducted using Statistical Package for the Social Sciences (SPSS) V.24.0 or higher.

REFERENCES:
- [Background] Prince MJ, Wu F, Guo Y, Gutierrez Robledo LM, O'Donnell M, Sullivan R, Yusuf S. The burden of disease in older people and implications for health policy and practice. Lancet. 2015 Feb 7;385(9967):549-62. doi: 10.1016/S0140-6736(14)61347-7. Epub 2014 Nov 6. PMID 25468153
- [Background] Murray SA, Firth A, Schneider N, Van den Eynden B, Gomez-Batiste X, Brogaard T, Villanueva T, Abela J, Eychmuller S, Mitchell G, Downing J, Sallnow L, van Rijswijk E, Barnard A, Lynch M, Fogen F, Moine S. Promoting palliative care in the community: production of the primary palliative care toolkit by the European Association of Palliative Care Taskforce in primary palliative care. Palliat Med. 2015 Feb;29(2):101-11. doi: 10.1177/0269216314545006. Epub 2014 Nov 13. PMID 25395577
- [Background] Mitchell GK. How well do general practitioners deliver palliative care? A systematic review. Palliat Med. 2002 Nov;16(6):457-64. doi: 10.1191/0269216302pm573oa. PMID 12465692
- [Background] McWhinney IR, Stewart MA. Home care of dying patients. Family physicians' experience with a palliative care support team. Can Fam Physician. 1994 Feb;40:240-6. PMID 7510562
- [Background] Morrison RS, Dietrich J, Ladwig S, Quill T, Sacco J, Tangeman J, Meier DE. Palliative care consultation teams cut hospital costs for Medicaid beneficiaries. Health Aff (Millwood). 2011 Mar;30(3):454-63. doi: 10.1377/hlthaff.2010.0929. PMID 21383364
- [Background] Hall S, Kolliakou A, Petkova H, Froggatt K, Higginson IJ. Interventions for improving palliative care for older people living in nursing care homes. Cochrane Database Syst Rev. 2011 Mar 16;2011(3):CD007132. doi: 10.1002/14651858.CD007132.pub2. PMID 21412898
- [Background] De Korte-Verhoef MC, Pasman HR, Schweitzer BP, Francke AL, Onwuteaka-Philipsen BD, Deliens L. General practitioners' perspectives on the avoidability of hospitalizations at the end of life: A mixed-method study. Palliat Med. 2014 Jul;28(7):949-958. doi: 10.1177/0269216314528742. Epub 2014 Apr 2. PMID 24694377
- [Background] Beernaert K, Deliens L, De Vleminck A, Devroey D, Pardon K, Van den Block L, Cohen J. Is There a Need for Early Palliative Care in Patients With Life-Limiting Illnesses? Interview Study With Patients About Experienced Care Needs From Diagnosis Onward. Am J Hosp Palliat Care. 2016 Jun;33(5):489-97. doi: 10.1177/1049909115577352. Epub 2015 Apr 7. PMID 25852203
- [Background] K, T. Using prognostic indicator guidance to plan care for final stages of life. Prim. Heal. Care 6, 25-28 (2010).
- [Background] Abarshi EA, Echteld MA, Van den Block L, Donker GA, Deliens L, Onwuteaka-Philipsen BD. Recognising patients who will die in the near future: a nationwide study via the Dutch Sentinel Network of GPs. Br J Gen Pract. 2011 Jun;61(587):e371-8. doi: 10.3399/bjgp11X578052. PMID 21801517
- [Background] Maas EA, Murray SA, Engels Y, Campbell C. What tools are available to identify patients with palliative care needs in primary care: a systematic literature review and survey of European practice. BMJ Support Palliat Care. 2013 Dec;3(4):444-51. doi: 10.1136/bmjspcare-2013-000527. PMID 24950525
- [Background] Walsh RI, Mitchell G, Francis L, van Driel ML. What Diagnostic Tools Exist for the Early Identification of Palliative Care Patients in General Practice? A systematic review. J Palliat Care. 2015;31(2):118-23. doi: 10.1177/082585971503100208. No abstract available. PMID 26201214
- [Background] Hamano J, Oishi A, Kizawa Y. Prevalence and Characteristics of Patients Being at Risk of Deteriorating and Dying in Primary Care. J Pain Symptom Manage. 2019 Feb;57(2):266-272.e1. doi: 10.1016/j.jpainsymman.2018.11.006. Epub 2018 Nov 15. PMID 30447382
- [Background] Gomez-Batiste X, Martinez-Munoz M, Blay C, Amblas J, Vila L, Costa X, Espaulella J, Espinosa J, Constante C, Mitchell GK. Prevalence and characteristics of patients with advanced chronic conditions in need of palliative care in the general population: a cross-sectional study. Palliat Med. 2014 Apr;28(4):302-11. doi: 10.1177/0269216313518266. Epub 2014 Jan 8. PMID 24403380
- [Background] Highet G, Crawford D, Murray SA, Boyd K. Development and evaluation of the Supportive and Palliative Care Indicators Tool (SPICT): a mixed-methods study. BMJ Support Palliat Care. 2014 Sep;4(3):285-90. doi: 10.1136/bmjspcare-2013-000488. Epub 2013 Jul 25. PMID 24644193
- [Background] Cohen J. A power primer. Psychol Bull. 1992 Jul;112(1):155-9. doi: 10.1037//0033-2909.112.1.155. PMID 19565683
- [Background] Hamano J, Oishi A, Kizawa Y. Identified Palliative Care Approach Needs with SPICT in Family Practice: A Preliminary Observational Study. J Palliat Med. 2018 Jul;21(7):992-998. doi: 10.1089/jpm.2017.0491. Epub 2018 Feb 9. PMID 29425053
- [Background] Pimentel, J. P., Durval, M., Araújo, F. O. & Guerreiro, A. C. ACeS Baixo Mondego. (2017).
- [Background] Martin Rosello ́ ML, Fernandez Lopez A, Sanz-Amores R, et al. Instrument Diagnosing Complexity in Palliative Care, IDC-Pal. Junta Andaluc ́ıa Cons Igualdad, Salud y Pol ́ıticas Soc [Internet] 2014. Available from: http://www.juntadeandalucia.es/salud/export/sites/csalud/galerias/documentos/ p_3_p_3_procesos_asistenciales_integrados/cuidados_paliativos/idc_pal_ 2014.pdf. [Accessed 6 April 2019].

DOCUMENTS (1):
  • Study Protocol (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT04010136/Prot_000.pdf